CLINICAL TRIAL: NCT02867267
Title: The Efficacy and Safety of Thymosin Alpha 1 for Sepsis: a Multicenter , Double-Blinded, Randomized and Controlled Clinical Trial
Brief Title: The Efficacy and Safety of Ta1 for Sepsis
Acronym: TESTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: SciClone Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Wu Jianfeng, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDX-2015-11
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Sepsis
Keywords: thymosin alpha 1; thymalfasin; sepsis; immunodepression
MeSH Terms: conditions — Sepsis | interventions — Thymalfasin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thymosin alpha 1 (Experimental): 1ml subcutaneous injection with 1.6 mg thymosin alpha 1, every 12±2 hours for not more than 7 days depending on the change of the subjects' condition
  Interventions: Drug: Thymosin alpha 1
- Placebo (Placebo Comparator): 1ml subcutaneous injection with placebo, every 12±2 hours for not more than 7 days depending on the change of the subjects' condition
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Thymosin alpha 1 — Subcutaneous injections of 1.6 mg thymosin alpha 1 every 12±2 hours for not more than 7 days depending on the change of the subjects' condition, prior to administration, the lyophilized powder is to be reconstituted with 1 ml of the provided diluent.
  Other Names: thymalfasin
  Arms: thymosin alpha 1
Other: Placebo — Subcutaneous injections of placebo every 12±2 hours for not more than 7 days depending on the change of the subjects' condition, prior to administration, the lyophilized powder is to be reconstituted with 1 ml of the provided diluent.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether thymalfasin is safe and effective in patients who have sepsis

DETAILED DESCRIPTION:
Our previous study reported that the 7-day treatment of Ta 1 demonstrated positive active effect as to the 28-day all-cause mortality and the augmentation of mHLA-DR (monocyte Human Leukocyte Antigen DR) at the secondary endpoint. Therefore, we intend to verify this finding through a randomized, double-blind and placebo-controlled clinical trial and the trail will include subjects with impaired immunologic functions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤85;
2. Signed informed consent signed;
3. Diagnosed as a sepsis according to the sepsis diagnosis criteria in "Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016": at least one acute severe organ dysfunction related to sepsis, and total SOFA scores ≥2;
4. Infected focus are confirmed or suspected and satisfy at least one of the followings:

   1. pathogenic microbes grow in blood or at aseptic locations
   2. presence of abscess or partially-infected tissues
   3. suspected infection identified by at least one of the following evidences:

      * leukocytes at normal aseptic locations
      * organic perforation (confirmed by imaging evidence, examination result or intestinal content leak during drainage)
      * Imaging evidence of pneumonia accompanied by purulent secretion
      * Related syndromes with high infection risk (cholangitis for example)

Exclusion Criteria:

1. History of organ or bone marrow transplantation;
2. Acute phase connective tissue diseases (such as rheumatoid diseases, systemic lupus erythematosus) and glomerulonephritis;
3. Under pregnancy or in suckling period;
4. Presence of hematologic malignancies;
5. The patient has received radiotherapy or chemotherapy within the past 30 days;
6. The patient is inclined to stop or cancel the artificial intervention for sustaining life, in other words, has abandoned treatment;
7. The patient has in the past 30 days received immunosuppressive drugs (tripterygium wilfordii, CellCept, cyclophosphamide, FK506, etc.) or received continuous treatment with prednisolone >10 mg/day (or the same dose of other hormones);
8. The patient could die of an underlying disease within 28 days or is in end-stage;
9. The patient has undergone CPR in the 72 hours before signing the informed consent and the neuromechanism has not fully recovered (GCS score ≤ 8);
10. The patient has in the past 30 days used thymosin or undergone certain clinical drug or instrument trials which could affect immunity (such as Xuebijing, ulinastatin and CRRT);
11. The patient has a medical history of allergy or intolerance to thymalfasin;
12. The source of infection cannot be contained, for example: infections that cannot be handled during surgical operations and drainage.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1106 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
28-day all-cause mortality | 28 days

SECONDARY OUTCOMES:
Incidence of new onset infection within 28 days | 28 days
  from initial injection on day 0 to day 28
28-day clearance rate of pathogenic microorganism | 28 days
ICU stays | 90 days
Hospital stays | 28 days
28-day re-hospitalization rate | 28 days
Changes of SOFA score at screening, end of CTM, days 7 (if applicable), day 14 and day 28 | 28 days
90-day all-cause mortality | 90 days
ICU mortality | 90 days
Ventilator-free days within 28 days | 28 days
ICU-free days within 28 days | 28 days
CRRT-free days within 28 days | 28 days
Vasoactive agents-free days within 28 days | 28 days
90-day SF-36 QOL scale | 90 days
Variance of the count of monocyte human lymphocyte antigens-DR (mHLA-DR) at days 7, 14 and 28 compared with the baseline at screening | 28 days
The percentage of Treg cells at screening and days 7 | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Guan Xiangdong, M. D, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (22):
- China (22):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing General Hospital of Nanjing Military Commend, Nanjing, Jiangsu
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu J, Zhou L, Liu J, Ma G, Kou Q, He Z, Chen J, Ou-Yang B, Chen M, Li Y, Wu X, Gu B, Chen L, Zou Z, Qiang X, Chen Y, Lin A, Zhang G, Guan X. The efficacy of thymosin alpha 1 for severe sepsis (ETASS): a multicenter, single-blind, randomized and controlled trial. Crit Care. 2013 Jan 17;17(1):R8. doi: 10.1186/cc11932. PMID 23327199
- [Result] Romani L, Bistoni F, Montagnoli C, Gaziano R, Bozza S, Bonifazi P, Zelante T, Moretti S, Rasi G, Garaci E, Puccetti P. Thymosin alpha1: an endogenous regulator of inflammation, immunity, and tolerance. Ann N Y Acad Sci. 2007 Sep;1112:326-38. doi: 10.1196/annals.1415.002. Epub 2007 May 10. PMID 17495242
- [Result] Romani L, Moretti S, Fallarino F, Bozza S, Ruggeri L, Casagrande A, Aversa F, Bistoni F, Velardi A, Garaci E. Jack of all trades: thymosin alpha1 and its pleiotropy. Ann N Y Acad Sci. 2012 Oct;1269:1-6. doi: 10.1111/j.1749-6632.2012.06716.x. PMID 23045964
- [Result] Wang X, Li W, Niu C, Pan L, Li N, Li J. Thymosin alpha 1 is associated with improved cellular immunity and reduced infection rate in severe acute pancreatitis patients in a double-blind randomized control study. Inflammation. 2011 Jun;34(3):198-202. doi: 10.1007/s10753-010-9224-1. PMID 20549321
- [Derived] Wu J, Pei F, Zhou L, Li W, Sun R, Li Y, Wang Z, He Z, Zhang X, Jin X, Long Y, Cui W, Wang C, Chen E, Zeng J, Yan J, Lin Q, Zhou F, Huang L, Shang Y, Duan M, Zheng W, Zhu D, Kou Q, Zhang S, Liu Y, Yao C, Shang M, Peng S, Zhou Q, Cheng KK, Guan X; TESTS study collaborator group. The efficacy and safety of thymosin alpha1 for sepsis (TESTS): multicentre, double blinded, randomised, placebo controlled, phase 3 trial. BMJ. 2025 Jan 15;388:e082583. doi: 10.1136/bmj-2024-082583. PMID 39814420